CLINICAL TRIAL: NCT06776848
Title: A Pilot, Multicentre, Controlled, Open-label Study Evaluating 24 Months of Lithium Carbonate Treatment in Patients With TBR1-related Neurocognitive Disorder
Acronym: ESALIT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAMBOT PHRCN 2021
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Proven Pathogenic or Probably Pathogenic TBR1 Variant
MeSH Terms: interventions — Biological Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groupe A (Experimental)
  Interventions: Other: Observation phase; Drug: Lithium treatment; Biological: biological monitoring
- Groupe B (Experimental)
  Interventions: Other: Observation phase; Drug: Lithium treatment; Biological: biological monitoring

INTERVENTIONS:
Other: Observation phase — Start of the observation phase for all patients for a period of 6 months. Group B: continuation of the observation phase for a further 6 months
Drug: Lithium treatment — The daily dose of lithium will be increased until the target lithiaemia is reached, while monitoring tolerance and possible adverse effects.
Biological: biological monitoring — The blood level of lithium will be monitored by regular blood tests
  - every 4 days until a targeted blood level is obtained

SUMMARY:
TBR1 is a human gene encoding a brain-specific transcription factor, principally expressed in the excitatory neurons of the neocortex. It regulates development of axonal projection and expression of numerous genes involved in autism spectrum disorders (ASD) and intellectual disability (ID). Recent progress in detection and analysis of rare variants allowed to identify group of genes with strong statistical evidence for association with ASD risk, of which TBR1. Numerous studies on mice showed that TBR1 heterozygous mice display autistic traits as deficiencies in social interaction, in cognitive flexibility, and in associative memory. Functional analyses on human cell lines have demonstrated that de novo truncating variants in TBR1 identified in patients with sporadic ASD disrupt transcriptional repression activity, localization, homodimerization of TBR1 product.

In 2019, only 12 single nucleotide variants (SNVs) and few copy number variations (CNVs) involving TBR1 have been reported in the literature and clinical descriptions were poor. To provide details on the phenotype linked to TBR1 mutations, we and others gathered 25 new individuals with de novo TBR1 SNV and CNV, complemented by a review of individuals previously reported in the literature. On 38 individuals, all presented developmental delay (DD)/ID, ranging from mild to severe, and 76% of them presented autistic traits. Additional behaviour disorders were observed in 85% of individuals, mainly attention deficit and aggressive behaviour. However, the natural history of patients with TBR1 variations is not well known.

Development of RNA-Seq allowed a better understanding of its transcription factor role and revealed that Tbr1 promotes expression of layer 6 markers as Wnt7b. In heterozygous and homozygous TBR1 mutant mice, Fazel Darbandi et al (1), observed that Wnt7b expression is reduced in cortical layer 6 and that neurons have reduced excitatory and inhibitory synaptic density. They showed that lithium chloride and lithium carbonate, WNT-signalling agonists, rescue the dendritic spines, the synaptic and the axonal defects in Tbr1layer5, Tbr1layer6 and Tbr1 constitutive (Tbr1+/-) mutant mice. They also observed an improvement of social interactions in mice after treatment by lithium. These results suggest an important and novel biological mechanism underlying ASD that may have implications for the treatment of patients with TBR1 variants.

Moreover, lithium treatment has already been evaluated in patients with neurocognitive disorders not linked to TBR1 showing an improvement in the adaptative behaviour and cognition function.

As of today, only symptomatic treatments are available. As lithium increase neuronal activity in mice, and may thus improve the symptoms of this disorder, we propose a clinical trial to study the security and efficacy of lithium carbonate targeting the patients with TBR1-related disorders, with specific and adapted endpoints. Lithium carbonate treatment will be administered after an observation period of 6 to 12 months, allowing to ascertain the stability of neurocognitive abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient, parent or legal representative
* ≥6 years old at the time of consent
* Proven pathogenic or probably pathogenic TBR1 variant (SNV confirmed by Sanger sequencing or CNV including only TBR1)
* If applicable: Stable concomitant psychoactive medication regimen (dose and schedule) ≥2 months prior to lithium initiation
* Affected individuals able to take tablet /capsules orally
* Highly effective method of contraception in affected female individuals of childbearing age (Combined hormonal contraception, progestogen-only hormonal contraception, intrauterine device, intrauterine hormone-releasing system) during treatment and for at least 3 months after the final dose of lithium
* Highly effective method of contraception in affected men individuals of childbearing age (condom) during the treatment and for at least 5 days after the final dose of lithium
* 1 available parent/guardian able to attend all visits having acceptable reading skills

Exclusion Criteria:

Criteria related to associated pathologies leading to particular risks:

* Renal/liver insufficiency (disturbed liver function, abnormal creatinine clearance)
* Unbalanced thyroid or diabetic pathology
* Long QT/Brugada syndrome or familial antecedent of Brugada syndrome, cardiac insufficiency
* Addison disease, dehydration, sodium restriction
* Non-stabilized epileptic disease.

Criteria related to contra-indication to treatment:

* Patient with concomitant diseases for which the experimental treatment by lithium could alter the tolerance
* Hypersensitivity to lactose, lithium or one of its excipients
* Patient with a wheat allergy (other than celiac disease)
* Pregnant or breastfeeding woman

Criteria related to treatments/procedures:

* Parent/guardian incapable of expressing consent
* Person not affiliated to a national health insurance scheme
* Person subject to a court order
* Cognitivo-behavioural therapy focused on ASD in 6 weeks previous to inclusion
* Other genetic pathogenic variant associated to neurocognitive disorders
* Any introduction of psychotropic molecules within 2 months prior to the trial, including neuroleptics, monoamine oxidase inhibitors, stimulants, antidepressants.
* Concomitant use of Angiotensin-Converting Enzyme (ACE) inhibitor, angiotensin II receptor antagonists, Nonsteroidal anti-inflammatory drugs, diuretics.
* Current lithium treatment
* Severe behavioural disorder or refusal to take drug treatment not allowing for compliance with medication;
* Impossibility to perform blood tests to check the lithiaemia when the patient is included.
* Participation in another therapeutic trial

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2027-09-12 (Estimated); Study Completion 2027-09-12 (Estimated)

PRIMARY OUTCOMES:
improvement in the Vineland II Adaptive Behaviour Scale (VABS-II) score ≥ standard error of the mean of the VABS-II | at the end of the 24 months of lithium carbonate treatment compared to baseline (end of the observational period)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France